CLINICAL TRIAL: NCT04171219
Title: A Phase 2 Basket Study of BXCL701, a Small Molecule Inhibitor of Dipeptidyl Peptidases (DPP), Administered in Combination With Pembrolizumab in Patients With Advanced Solid Cancers
Brief Title: Talabostat and Pembrolizumab for the Treatment of Advanced Solid Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: There is no PR/CR observed in the first stage, so study stopped without proceeding to the stage 2 of efficacy stage.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0748; NCI-2019-07569 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0748 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Advanced Malignant Solid Neoplasm; Recurrent Malignant Solid Neoplasm
MeSH Terms: interventions — pembrolizumab; PT-100 dipeptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (talabostat, pembrolizumab) (Experimental): Patients receive talabostat PO BID on days 1-14 and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Talabostat Mesylate

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Talabostat Mesylate — Given PO
  Other Names: Val-boro-Pro

SUMMARY:
This phase II trial studies the side effects of talabostat and pembrolizumab and to see how well they work for the treatment of solid cancers that have spread to other places in the body (advanced). Talabostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving talabostat and pembrolizumab may help control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate response rate per Response Evaluation Criteria in Solid Tumors (RECIST) and immune (i)RECIST in patients treated in cohort A and in patients treated in cohort B.

II. To evaluate dose-limiting toxicities (DLT) in the first 6 patients enrolled to the study.

SECONDARY OBJECTIVES:

I. To evaluate progression-free survival (PFS). II. To evaluate duration of response (DOR). III. To evaluate overall survival (OS). IV. To evaluate overall safety and tolerability.

EXPLORATORY OBJECTIVES:

I. To evaluate the quantitative and qualitative effects of talabostat (BXCL701) in combination with pembrolizumab on relevant immune effector cytokines in blood.

II. To evaluate the quantitative and qualitative effects of BXCL701 in combination with pembrolizumab on various immunological effector cells, including neutrophils, myeloid derived suppressor cells (MDSCs), dendritic cells, cancer associated fibroblast (CAF), T-cells and macrophage density in pre-dose tumor biopsies and when feasible in post-dose tumor tissues.

III. To explore the predictive value of baseline programmed death ligand 1 (PD-L1) tumor expression and tumor mutation burden (TMB) with clinical outcomes.

IV. To evaluate changes in serially collected blood circulating tumor deoxyribonucleic acid (DNA) (ctDNA) to assess for tumor response and clonal evolution.

V. To evaluate pre- and post-treatment PD-L1 positron emission tomography (PET)/computed tomography (CT) as a predictive tool for therapeutic efficacy.

OUTLINE:

Patients receive talabostat orally (PO) twice daily (BID) on days 1-14 and pembrolizumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a histology or cytology proven solid advanced cancer, which failed or is intolerant of standard therapies known to offer survival benefit unless standard therapies include PD1 or PD-L1 antibodies

  * Lead-in stage: patient with advanced cancers meeting the criteria above with or without prior treatment with PD1/PDL1 antibodies. Patients with prior treatment with PD1/PDL1 antibodies should be relapsed
  * Efficacy stage cohort A: patients with advanced cancers not previously treated with PD1/PDL1 antibodies
  * Efficacy stage cohort B: patients with advanced cancers which have relapsed or progressed with PD1/PDL1 antibodies
* Patient with a life expectancy of more than 3 months, in the opinion of the investigator
* Patient has Eastern Cooperative Oncology Group (ECOG) performance status of 0 2
* Patients < 18 years of age have to weigh > 40 kgs
* Patients must have measurable disease by RECIST 1.1 and iRECIST. Disease amenable to a biopsy is not mandatory
* Patient's acute toxic effects of previous anticancer therapy have resolved to =< grade 1 except for grade 2 peripheral neuropathy or any grade of alopecia
* Serum creatinine =< 1.5 times institutional upper limit of normal (ULN) or calculated creatinine clearance > 40 mL/min
* Serum albumin >= 2.5 g/dL
* Total bilirubin =< 1.5 x ULN (for patients with known Gilbert syndrome < 3 x ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x institutional ULN (patients with hepatic metastases must have AST/ALT =< 5 x ULN)
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* Hemoglobin >= 8 g/dL and no red blood cell transfusions during the prior 7 days
* Platelet count >= 75 x 10^9/L
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 14 days prior to the initiation of treatment and/or postmenopausal women must be amenorrhoeic for at least 12 months to be considered of non-childbearing potential. Women of childbearing potential must agree and commit to the use of 2 highly effective methods of birth control throughout the duration of the study until at least 4 months following the last dose of study drug. Acceptable methods are defined as those that result, alone or in combination, in a low failure rate (ie, less than 1% per year) when used consistently and correctly, such as surgical sterilization, an intrauterine device, or hormonal contraception in combination with a barrier method. It is currently unknown whether BXCL701 or pembrolizumab may reduce the effectiveness of systemically acting hormonal contraceptives; therefore, women using systemically acting hormonal contraceptives should add a barrier method. In certain countries (if permitted by law), WOCBP may agree to abide by heterosexual sexual abstinence during the time of participation in this study
* Male patients and their female partners of childbearing potential must agree and commit to use a barrier contraception (eg, condom with spermicidal foam/gel/film/cream/suppository) throughout the duration of the study until at least 60 days following the last dose of study drug, in addition to their female partners using either an intrauterine device or hormonal contraception and continuing until at least 4 months days following the last dose of study drug. This criterion may be waived for male patients who have had a vasectomy > 6 months before signing the informed consent form (ICF)
* Patient has signed informed consent prior to initiation of any study-specific procedures or treatment
* Patient is able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Patient cannot swallow oral medication
* Patient is on gliptins
* Patient has active central nervous system (CNS) metastases not controlled by prior surgery or radiotherapy (patient must be off steroids). Patients with signs or symptoms suggestive of brain metastasis are not eligible unless brain metastases are ruled out by brain magnetic resonance imaging/computed tomography (MRI/CT)
* Patient has received external-beam radiation or another systemic anticancer therapy within 14 days or 5 half-lives, whichever is shorter, prior to study treatment
* Patient has received treatment with an investigational systemic anticancer agent within 14 days prior to study drug administration
* Patient has an additional active malignancy that may confound the assessment of the study endpoints. Patients with the following concomitant neoplastic diagnoses are eligible: non-melanoma skin cancer and carcinoma in situ (including transitional cell carcinoma, anal carcinoma, and melanoma in situ). Patients with simultaneous cancers, which are not active and do not require treatment may be eligible contingent on discussion with the principle investigator (PI) and supporter
* Patient has clinically significant cardiovascular disease (e.g., uncontrolled or any New York Heart Association class 3 or 4 congestive heart failure, uncontrolled angina, history of myocardial infarction, unstable angina or stroke within 6 months prior to study entry, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication)
* Patient has a diagnosis of immunodeficiency or is receiving systemic steroid therapy at a prednisone equivalent dose of > 10 mg daily for at least 1 week or other form of immunosuppressive therapy within 7 days prior to cycle 1 day 1 (C1D1)
* Patient has uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, disseminated intravascular coagulation, or psychiatric illness/social situations that would limit compliance with study requirements
* Patient has known positive status for human immunodeficiency virus active or chronic hepatitis B or hepatitis C. Patients with history of hepatitis B or C and undetectable viral load are eligible. Screening is not required
* Has a clinically significant upper gastrointestinal obstruction, abnormal physiological function or malabsorption syndrome that may affect the absorption of the study medication
* Patient has any medical condition which, in the opinion of the investigator, places the patient at an unacceptably high risk for toxicity
* Patient is pregnant or breast-feeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an open-label, single-institution, Phase 2 study of BXCL701 administered orally and daily, combined with pembrolizumab, in PD1/PDL1 or CTLA-4 naïve and PD1/PDL1 or CTLA-4 pretreated patients with advanced solid cancers at The University of Texas MD Anderson Cancer Center.
Groups:
- Cohort A: PD-1/PD-L1 and/or CTLA-4 Inhibitor Treatment naïve; Cohort B: PD-1/PD-L1 and/or CTLA-4 Inhibitor Pretreated: BXCL701: 0.3 mg orally twice a day on Days 1 to 14 of a 21-day cycle plus pembrolizumab 200 mg administered IV on Day 1 every 21 days
Period: Overall Study
Arm/Group | Cohort A: PD-1/PD-L1 and/or CTLA-4 Inhibitor Treatment naïve | Cohort B: PD-1/PD-L1 and/or CTLA-4 Inhibitor Pretreated
Started | 14 | 17
Completed | 0 | 0
Not Completed | 14 | 17
Not completed — Adverse Event | 1 | 0
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 9 | 13
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Clinical PD and extended treatment holding/ Patient choice/withdrew consent | 1 | 1
Not completed — Clinical PD/Patient choice | 1 | 0
Not completed — Toxicity/ Patient choice | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: PD-1/PD-L1 and/or CTLA-4 Inhibitor Treatment naïve | Cohort B: PD-1/PD-L1 and/or CTLA-4 Inhibitor Pretreated | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 13 | 20
  >=65 years | 7 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 9 | 12 | 21
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 17 | 31

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate Per RECIST v1.1
Description: Disease control rate was defined as the percentage of patients who had complete response (CR), partial response (PR), or stable disease (SD) according to RECIST v1.1.
Time Frame: At baseline and at the end of Cycle 3 (approximately 9 weeks after the first study treatment dose), and then approximately every 9 weeks thereafter until development of progressive disease, up to 3 years
Population: To be evaluable for response, patients must have completed at least 9 weeks of treatment and received at least 70% of the total planned talabostat dose in cycles 1 and 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: PD-1/PD-L1 and/or CTLA-4 Inhibitor Treatment naïve | Cohort B: PD-1/PD-L1 and/or CTLA-4 Inhibitor Pretreated
Number analyzed (Participants) | 9 | 10
Participants | 4 | 4

2. Primary Outcome: Immune-related Disease Control Rate Per iRECIST
Description: Immune-related disease control rate was defined as the percentage of patients who had immune-related complete response (iCR), immune-related partial response (iPR), or immune-related stable disease (iSD) according to iRECIST.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: PD-1/PD-L1 and/or CTLA-4 Inhibitor Treatment naïve | Cohort B: PD-1/PD-L1 and/or CTLA-4 Inhibitor Pretreated
Number analyzed (Participants) | 9 | 10
Participants | 4 | 5

3. Primary Outcome: Dose-limiting Toxicities (DLTs)
Description: A DLT was defined as any of the following AEs occurring during Cycle 1, regardless of investigator attribution to study treatment:
  * Any Grade 4 laboratory abnormality, regardless of duration.
  * Any Grade 3 laboratory abnormalities if associated with clinical symptoms regardless of duration
  * Any Grade ≥3 non-hematologic AE, with the exceptions of Grade ≥3 nausea, vomiting, diarrhea, constipation, and fatigue, that resolves to Grade ≤1 within 72 hours with optimal medical management and/or supportive measures.
  * Grade ≥3 thrombocytopenia with Grade >1 bleeding or requirement for platelet transfusion.
  * Grade ≥3 febrile neutropenia.
  * Grade ≥3 fever.
  * Grade ≥3 skin rash.
  * AST or ALT >3 × upper limit of normal [ULN] with concomitant total bilirubin >2 × ULN.
  * Any toxicity resulting in ≥30% held/skipped doses of BXCL701 during Cycle 1.
  * Delay of Cycle 2 by ≥14 days due to toxicity.
  * Any other significant toxicity considered by the investigatoro be dose-limiting.
Time Frame: DLT was assessed during Cycle 1 (21-day cycle)
Population: DLT was assessed in the first 6 patients enrolled on the study. Unless doses were held because of DLT, a patient must have received >70% of their BXCL701 in Cycle 1 (i.e., ≥30 of 42 planned doses) with pembrolizumab dosed on Day 1 of Cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: PD-1/PD-L1 and/or CTLA-4 Inhibitor Treatment naïve | Cohort B: PD-1/PD-L1 and/or CTLA-4 Inhibitor Pretreated
Number analyzed (Participants) | 2 | 4
Participants | 1 | 0

4. Secondary Outcome: Progression-free Survival (PFS) by RECIST v1.1
Description: PFS was defined as the time from administration of the first dose to the first documented disease progression by RECIST v1.1 or death due to any cause, whichever occurs first. Patients who were alive and had not experienced disease progression at the time of data cutoff were censored.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: PD-1/PD-L1 and/or CTLA-4 Inhibitor Treatment naïve | Cohort B: PD-1/PD-L1 and/or CTLA-4 Inhibitor Pretreated
Number analyzed (Participants) | 9 | 10
Months | 2.7 [1.9 to 7.8] | 2.5 [2.1 to 6.5]

5. Secondary Outcome: Progression-free Survival (PFS) by iRECIST
Description: PFS was defined as the time from administration of the first dose to the first documented disease progression by iRECIST v1.1 or death due to any cause, whichever occurs first. Patients who were alive and had not experienced disease progression at the time of data cutoff were censored.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: PD-1/PD-L1 and/or CTLA-4 Inhibitor Treatment naïve | Cohort B: PD-1/PD-L1 and/or CTLA-4 Inhibitor Pretreated
Number analyzed (Participants) | 9 | 10
Months | 2.7 [1.9 to 7.8] | 2.5 [2.1 to 6.5]

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was measured from the first date of administration of the study drug to the date of death due to any cause. Patients who were alive at the last follow-up examination were censored.
Time Frame: From the first date of administration of the study drug to the date of data cut-off (January 7, 2024)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: PD-1/PD-L1 and/or CTLA-4 Inhibitor Treatment naïve | Cohort B: PD-1/PD-L1 and/or CTLA-4 Inhibitor Pretreated
Number analyzed (Participants) | 9 | 10
Months | 16.4 [4.4 to 30.1] | 26.1 [8.6 to NA] — not estimated

7. Secondary Outcome: Treatment-related Adverse Event (TRAE)
Description: All safety data from all patients, who received at least one dose of study drug were included in safety analysis. Each AE (as defined by NCI CTCAE v5) was counted only once for a given subject. In the event a patient experienced repeated episodes of the same AE, then the event with the highest severity and/or strongest causal relationship to study treatment was used for purposes of tabulations.
Time Frame: Patients were monitored for AE from the first day of administration of study medication through 30 days following the last dose of BXCL701 and or pembrolizumab, an average of 3 years.
Population: All patients who received at least one dose of study drug were included in safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: PD-1/PD-L1 and/or CTLA-4 Inhibitor Treatment naïve | Cohort B: PD-1/PD-L1 and/or CTLA-4 Inhibitor Pretreated
Number analyzed (Participants) | 14 | 17
Participants | 10 | 9

ADVERSE EVENTS:
Time Frame: Patients were monitored for AE from the first day of administration of study medication through 30 days following the last dose of BXCL701 and or pembrolizumab, an average of 3 years.
Description: All AEs were reported to regulatory authorities and investigators in accordance with all applicable regulations. AEs were graded per NCI CTCAE v4.03. Every attempt was made to report all SAEs to the IND Office, within 5 working days and all life-threatening or fatal events, unexpected and drug-related within 24 hours of knowledge of the event to the Safety Project Manager in the IND Office. Percentages are calculated using the number of patients in the safety population as the denominator.
Groups:
- All Patients Treated on This Study.: BXCL701: 0.3 mg orally twice a day on Days 1 to 14 of a 21-day cycle plus pembrolizumab 200 mg administered IV on Day 1 every 21 days
Arm/Group | All Patients Treated on This Study.
All-Cause Mortality (participants affected / at risk) | 26/31
Serious Adverse Events (participants affected / at risk) | 17/31
Other Adverse Events (participants affected / at risk) | 29/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Treated on This Study. (N=31)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Hypotension (Vascular disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Vulval infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Treated on This Study. (N=31)
Hypotension (Vascular disorders) | 8 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pain (General disorders) | 7 (7)
Fatigue (General disorders) | 6 (6)
General disorders and administration site conditions - Other, specify (General disorders) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Edema limbs (General disorders) | 4 (4)
Fever (General disorders) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypertension (Vascular disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Platelet count decreased (Investigations) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Lung infection (Infections and infestations) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Syncope (Nervous system disorders) | 2 (2)
White blood cell decreased (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Generalized edema (General disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vision decreased (Eye disorders) | 1 (1)
Vulval infection (Infections and infestations) | 1 (1)
Weight gain (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT04171219/Prot_SAP_002.pdf
  • Informed Consent Form (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT04171219/ICF_001.pdf